CLINICAL TRIAL: NCT03019640
Title: Immunotherapy With Ex Vivo-Expanded Cord Blood-Derived NK Cells Combined With Rituximab High-Dose Chemotherapy and Autologous Stem Cell Transplant for B-Cell Non-Hodgkin's Lymphoma
Brief Title: Umbilical Cord Blood NK Cells, Rituximab, High-Dose Chemotherapy, and Stem Cell Transplant in Treating Patients With Recurrent or Refractory B-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0751; NCI-2018-01239 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0751 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Results first posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-12

CONDITIONS: Mantle Cell Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Follicular Lymphoma; Recurrent Indolent Adult Non-Hodgkin Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Follicular Lymphoma; Refractory Indolent Adult Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — Carmustine; Cytarabine; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; Lenalidomide; Melphalan; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Treatment (chemotherapy, NK infusion, stem cell transplant) (Experimental): See Detailed Description.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carmustine; Biological: Cord Blood-derived Expanded Allogeneic Natural Killer Cells; Drug: Cytarabine; Drug: Etoposide; Biological: Filgrastim; Drug: Lenalidomide; Drug: Melphalan; Biological: Rituximab

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo stem cell transplant
  Other Names: Autologous Hematopoietic Cell Transplantation; autologous stem cell transplantation
Drug: Carmustine — Given IV
  Other Names: BCNU; Becenum; Becenun; BiCNU; Bis(chloroethyl) Nitrosourea; Bis-Chloronitrosourea; Carmubris; Carmustin; Carmustinum; FDA 0345; N,N''-Bis(2-chloroethyl)-N-nitrosourea; Nitrourean; Nitrumon; SK 27702; SRI 1720; WR-139021
Biological: Cord Blood-derived Expanded Allogeneic Natural Killer Cells — Given IV
  Other Names: Allogeneic CB-derived Ex vivo-expanded NK Cells; CB-derived Expanded Allogeneic NK Cells; UCB-derived Expanded Allogeneic NK Cells; Umbilical Cord Blood-derived Expanded Allogeneic Natural Killer Cells
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Biological: Filgrastim — Given SC
  Other Names: G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima

SUMMARY:
This phase II trial studies the side effects of cord blood-derived expanded allogeneic natural killer cells (umbilical cord blood natural killer [NK] cells), rituximab, high-dose chemotherapy, and stem cell transplant in treating patients with B-cell non-Hodgkin's lymphoma that has come back (recurrent) or that does not respond to treatment (refractory). Immune system cells, such as cord blood-derived expanded allogeneic natural killer cells, are made by the body to attack foreign or cancerous cells. Immunotherapy with rituximab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as carmustine, cytarabine, etoposide, lenalidomide, melphalan, and rituximab, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. A stem cell transplant using stem cells from the patient or a donor may be able to replace blood-forming cells that were destroyed by chemotherapy used to kill cancer cells. The donated stem cells may also replace the patient's immune cells and help destroy any remaining cancer cells. Giving cord blood-derived expanded allogeneic natural killer cells, rituximab, high-dose chemotherapy, and stem cell transplant may work better in treating patients with recurrent or refractory B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish the safety of this treatment by determining its treatment-related mortality (TRM) within 30 days.

SECONDARY OBJECTIVES:

I. To estimate the relapse-free survival (RFS). II. To estimate the overall survival (OS). III. To quantify duration of infused allogeneic umbilical cord blood (UCB)-derived natural killer (NK) cells in the recipient.

OUTLINE:

PREPARATIVE REGIMEN: Patients receive carmustine intravenously (IV) over 2 hours on day -12, etoposide IV twice daily (BID) over 3 hours on days -11 to -8, cytarabine IV BID over 1 hour on days -11 to -8, melphalan IV over 30 minutes on day -7, and lenalidomide orally (PO) once daily (QD) on days -7 to -2 in the absence of disease progression or unacceptable toxicity. Patients who are CD20+ also receive rituximab IV over 3 hours on days -13 and -7.

NK-CELL INFUSION: Patients receive cord blood-derived expanded allogeneic NK cells IV over 1 hour on day -5 in the absence of disease progression or unacceptable toxicity.

STEM CELL TRANSPLANT: Patients undergo stem cell transplant IV over 30-60 minutes on day 0 in the absence of disease progression or unacceptable toxicity.

POST-TRANSPLANT: Patients receive filgrastim subcutaneously (SC) QD beginning on day +5. Treatment continues until white blood cell count recovers in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30, 100, and 180 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with B-cell lymphoma who are candidates to autologous stem-cell transplantation:

  * Primary refractory or relapsed diffuse large B-cell lymphoma in response to salvage treatment
  * Primary refractory or relapsed follicular lymphoma or other indolent B-cell histology in response to salvage treatment
  * Chemosensitive mantle-cell lymphoma in first or later line of treatment
* Estimated serum creatinine clearance >= 60 ml/min and a normal serum creatinine for age
* Serum glutamic-oxaloacetic transaminase (SGOT) and/or serum glutamate pyruvate transaminase (SGPT) =< 3 x upper limit of normal (ULN)
* Total bilirubin and alkaline phosphatase (ALP) =< 2 x ULN or =< 3 x ULN for Gilbert's disease
* Forced expiratory volume in one second (FEV1), forced vital capacity (FVC) and diffusion lung capacity (DLCO) (corrected for hemoglobin [Hgb]) >= 50% of the predicted value
* Left ventricular ejection fraction >= 40%. No uncontrolled arrhythmias or symptomatic cardiac disease
* Performance status < 2 (Eastern Cooperative Oncology Group [ECOG])
* Negative beta human chorionic gonadotropin (HCG) in woman with child-bearing potential

Exclusion Criteria:

* Primary central nervous system (CNS) lymphoma
* Grade >= 3 non-hematologic toxicity from prior therapy that has not resolved to =< grade (G) 1
* Prior whole brain irradiation
* Active hepatitis B, either active carrier (hepatitis B surface antigen positive [HBsAg +]) or viremic (hepatitis B virus [HBV] deoxyribonucleic acid [DNA] >= 10,000 copies/mL, or >= 2,000 IU/mL)
* Evidence of either cirrhosis or stage 3-4 liver fibrosis in patients with chronic hepatitis C or positive hepatitis C serology
* Active infection requiring parenteral antibiotics
* Human immunodeficiency virus (HIV) infection
* Radiation therapy in the month prior to enroll
* Breastfeeding females

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yago L Nieto, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruitment from October 2017 to August 2021 at MD Anderson Cancer Center.
Groups:
- Treatment (Chemotherapy, NK Infusion, Stem Cell Transplant): Patients receive carmustine intravenously (IV) over 2 hours on day -12, etoposide IV twice daily (BID) over 3 hours on days -11 to -8, cytarabine IV BID over 1 hour on days -11 to -8, melphalan IV over 30 minutes on day -7, and lenalidomide orally (PO) once daily (QD) on days -7 to -2 in the absence of disease progression or unacceptable toxicity. Patients who are CD20+ also receive rituximab IV over 3 hours on days -13 and -7.
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, NK Infusion, Stem Cell Transplant)
Started | 22
Completed | 14
Not Completed | 8
Not completed — Screen Failures | 4
Not completed — Adverse Event | 3
Not completed — Participant Relapsed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy, NK Infusion, Stem Cell Transplant)
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Treatment-related Mortality Within 30 Days (TRM30)
Description: Participants that had Treatment-related mortality within 30 days.
Time Frame: Up to 30 days
Population: Four participants did not received treatment due to screen failures.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, NK Infusion, Stem Cell Transplant)
Number analyzed (Participants) | 18
Participants | 0

2. Secondary Outcome: Number of Participants Who Survived
Description: Number of Participants Who Survived at day 180.
Time Frame: From the time of transplant, assessed up to day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, NK Infusion, Stem Cell Transplant)
Number analyzed (Participants) | 22
Participants | 16

ADVERSE EVENTS:
Time Frame: All-Cause Mortality monitored/assessed up to 180 days.
Arm/Group | Treatment (Chemotherapy, NK Infusion, Stem Cell Transplant)
All-Cause Mortality (participants affected / at risk) | 2/22
Serious Adverse Events (participants affected / at risk) | 15/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Chemotherapy, NK Infusion, Stem Cell Transplant) (N=22)
Alanine aminotransferase increased (Hepatobiliary disorders) | 2
Anemia (Blood and lymphatic system disorders) | 1
Aspartate aminotransferase increased (Hepatobiliary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Cardiac disorders) | 1
Hypoxia (Hepatobiliary disorders) | 1
Infections and infestations (Infections and infestations) | 1
Lung (Infections and infestations) | 1
Lymphocyte count decreased (Blood and lymphatic system disorders) | 9
Neutrophil count decreased (Blood and lymphatic system disorders) | 12
Platelet count decreased (Blood and lymphatic system disorders) | 12
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
White blood cell decreased (Blood and lymphatic system disorders) | 15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Chemotherapy, NK Infusion, Stem Cell Transplant) (N=22)
Abdominal pain (General disorders) | 4
Acute kidney injury (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 10
Alkaline phosphatase increased (Investigations) | 6
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4
Anemia (Blood and lymphatic system disorders) | 22
Anorexia (Metabolism and nutrition disorders) | 13 — Anorexia
Anxiety (Psychiatric disorders) | 8
Arthralgia (Immune system disorders) | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Aspartate aminotransferase increased (Investigations) | 6
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Back pain (Injury, poisoning and procedural complications) | 2 — Back pain
Bladder infection (Infections and infestations) | 1
Bloating (Gastrointestinal disorders) | 3
Blood bilirubin increased (Investigations) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Chills (General disorders) | 7 — Chills
Cholesterol high (Investigations) | 2 — Cholesterol high
Constipation (Gastrointestinal disorders) | 12 — Constipation
Cough (General disorders) | 7 — Cough
Creatinine increased (Investigations) | 2 — Creatinine increased
Dehydration (Metabolism and nutrition disorders) | 4 — Dehydration
Diarrhea (Gastrointestinal disorders) | 21 — Diarrhea
Dizziness (Immune system disorders) | 9 — Dizziness
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 3 — Dyspepsia
Dysphagia (Gastrointestinal disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 — Dyspnea
Ear pain (Ear and labyrinth disorders) | 1 — Ear pain
Edema face (General disorders) | 1
Edema limbs (General disorders) | 12
Encephalopathy (Hepatobiliary disorders) | 1
Endocrine disorders (Endocrine disorders) | 1 — Endocrine disorders
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 5 — Esophagitis
Eye disorders (Eye disorders) | 1
Fatigue (General disorders) | 17
Febrile neutropenia (Blood and lymphatic system disorders) | 7
Fever (General disorders) | 22
Flatulence (Gastrointestinal disorders) | 1
Flushing (Immune system disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 — Gastroesophageal reflux disease
Gastrointestinal pain (Gastrointestinal disorders) | 1
General disorders and administration site conditions (General disorders) | 2 — General disorders and administration site conditions
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4
Headache (Nervous system disorders) | 11
Hematuria (Renal and urinary disorders) | 1 — Hematuria
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 18
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 2
Hypertension (Respiratory, thoracic and mediastinal disorders) | 7
Hyperuricemia (Metabolism and nutrition disorders) | 2 — Hyperuricemia
Hypoalbuminemia (Metabolism and nutrition disorders) | 10
Hypocalcemia (Metabolism and nutrition disorders) | 10
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 12
Hypotension (Vascular disorders) | 13 — Hypotension
Hypothyroidism (Endocrine disorders) | 1 — Hypothyroidism
Hypoxia (Investigations) | 4 — Hypoxia
Ileus (Gastrointestinal disorders) | 1 — Ileus
Immune system disorders (Immune system disorders) | 3
Infections and infestations (Infections and infestations) | 5
Infusion related reaction (General disorders) | 3
INR increased (Investigations) | 3
Insomnia (Psychiatric disorders) | 7 — Insomnia
Investigations (Investigations) | 7
Lung infection (Infections and infestations) | 1
Lymph node pain (Blood and lymphatic system disorders) | 1 — Lymph node pain
Lymphocyte count decreased (Investigations) | 22
Lymphocyte count increased (Investigations) | 1 — Lymphocyte count increased
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1
Mucosal infection (Infections and infestations) | 1 — Mucosal infection
Mucositis oral (Gastrointestinal disorders) | 17 — Mucositis oral
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 — Myalgia
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 — Nasal congestion
Nausea (Gastrointestinal disorders) | 22 — Nausea
Neck pain (Musculoskeletal and connective tissue disorders) | 1 — Neck pain
Nervous system disorders (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 22
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 6 — Pain
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 — Pain in extremity
Papulopustular rash (Infections and infestations) | 2 — Papulopustular rash
Paresthesia (Nervous system disorders) | 3 — Paresthesia
Peripheral motor neuropathy (Nervous system disorders) | 1 — Peripheral motor neuropathy
Platelet count decreased (Investigations) | 22 — Platelet count decreased
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 — Pleural effusion
Prostatic obstruction (Reproductive system and breast disorders) | 1 — Prostatic obstruction
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 — Pulmonary edema
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 — Rash acneiform
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 — Rash maculo-papular
Rectal pain (Gastrointestinal disorders) | 3 — Rectal pain
Renal and urinary disorders (Renal and urinary disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 — Respiratory failure
Restlessness (Nervous system disorders) | 1 — Restlessness
Sinus bradycardia (Cardiac disorders) | 1 — Sinus bradycardia
Sinus tachycardia (Cardiac disorders) | 14 — Sinus tachycardia
Sinusitis (Infections and infestations) | 1 — Sinusitis
Skin and subcutaneous tissue disorder (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 — Sore throat
Thromboembolic event (Vascular disorders) | 1
Tremor (Nervous system disorders) | 1
Upper respiratory infection (Infections and infestations) | 2
Urinary frequency (Renal and urinary disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Vascular disorders (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Weight gain (Investigations) | 1 — Weight gain
White blood cell decreased (Investigations) | 22 — White blood cell decreased

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/40/NCT03019640/Prot_SAP_000.pdf